CLINICAL TRIAL: NCT02825693
Title: The Development of Surgical Pathways Using Femto-second Laser Technology to Increase the Efficiency and Safety of Cataract Surgery Within a Public Health Sector Setting - A Randomised Controlled Trial
Brief Title: Femtosecond Laser Assisted Cataract Surgery in The NHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILH297-P002
Record Dates: First submitted 2016-06-20; First posted 2016-07-07 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-02

CONDITIONS: Cataract; Surgery
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

ARMS (2):
- Femtosecond laser cataract surgery (Active Comparator): Cataract surgery with femtosecond laser treatment for corneal incisions, astigmatic keratotomies, capsulotomy and nuclear fragmentation
  Interventions: Procedure: Femtosecond laser assisted cataract surgery
- Conventional phacoemulsification surgery (Active Comparator): Conventional phacoemulsification surgery
  Interventions: Procedure: Conventional cataract surgery (phacoemulsification)

INTERVENTIONS:
Procedure: Conventional cataract surgery (phacoemulsification)
  Arms: Conventional phacoemulsification surgery
Procedure: Femtosecond laser assisted cataract surgery
  Arms: Femtosecond laser cataract surgery

SUMMARY:
This study aims to examine the health economic impact of adopting femtosecond laser technology to assist high volume cataract surgery (FLACS) within a state-funded healthcare system, the National Health Service (NHS).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have reduced visual acuity or visual symptoms attributed to the presence of cataract in one or both eyes by the examining ophthalmologist or else must require cataract surgery on clinical grounds other than visual symptoms.
* Patients must be willing to attend for follow-up at 1 month after cataract surgery.
* Patients must be sufficiently fluent in English for informed consent and self-completion of the patient reported outcome questionnaires.

Exclusion Criteria:

* Children below the age of 18
* Already enrolled in another study

The principle exclusion criteria relate to clinical contraindications for FLACS, such as:

* Significant corneal opacities
* Small pupils following pharmacological dilatation
* Patients unable to lie sufficiently flat so as to be positioned underneath the laser machine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Cost-analysis: Healthcare resource use attributable to managing patients in this study will be collected. | up to 2 months
  These include (but not necessarily be limited to) the cost of surgery for both arms of the trial (including resource use and staffing levels required for the surgical protocols), resource use attributable to managing complications arising from surgery, all relevant diagnostic investigations, further surgery where necessary, hospital length of stay and ward type, outpatient attendances, procedures performed on an outpatient basis, Accident & Emergency attendances and prescribed drug medications. The quantity of resource use for each cost component will be measured from medical records. Site-specific unit costs will be taken in preference of standard published sources or national tariffs where possible.